CLINICAL TRIAL: NCT03388398
Title: Evaluation of the Population-level Impact of Prevention of Mother-to-Child HIV Transmission Program Option B+ in Zimbabwe
Brief Title: Evaluation of the Population-level Impact of PMTCT Option B+ in Zimbabwe
Status: Completed | Type: Observational
Sponsor: University of California, Berkeley (Other)
Collaborators: Centre for Sexual Health and HIV/AIDS Research Zimbabwe (CeSHHAR Zimbabwe) (Other); Consorcio de Investigación sobre VIH/SIDA/TB (CISIDAT). (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Liverpool School of Tropical Medicine (Other); Ministry of Health and Child Welfare, Zimbabwe (Other); Elizabeth Glaser Pediatric AIDS Foundation (Other); Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01HD080492-01 (NIH); 1R01HD080492-01 (NIH)
Record Dates: First submitted 2017-12-15; First posted 2018-01-03 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: HIV Infections
Keywords: Mother-to-child transmission of HIV (MTCT); Prevention of mother-to-child HIV transmission (PMTCT); Antiretroviral therapy (ART); Antenatal care (ANC); Pediatric infections; Pregnancy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spot samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Mother-Infant Pairs: Mothers or caregivers (at least 16 years of age) and their infants who are 9 to 18 months of age at the time of their survey.
- Mothers or caregivers: Mothers or caregivers (at least 16 years of age) who are 19 to 36 months postpartum at the time of the survey.
- Healthcare staff: Healthcare staff (employed staff and volunteers at least 18 years of age) at all participating healthcare facilities.
- Providers: Health care providers (at least 18 years of age) at select participating healthcare facilities.
- Patients: Patients (at least 18 years of age) receiving care at select participating healthcare facilities.

SUMMARY:
This study evaluates the impact of Zimbabwe's program for the prevention of mother-to-child HIV transmission (PMTCT) on vertical transmission of HIV infection and HIV-free survival among infants exposed to HIV. The study will test the hypothesis that the accelerated PMTCT program in Zimbabwe will result in fewer new HIV infections in infants and will increase infant survival.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends that all pregnant women receive antiretroviral therapy (ART) during pregnancy and breastfeeding ("Option B") or ideally throughout their lives regardless of clinical stage ("Option B+"). In February 2013, Zimbabwe's Ministry of Health and Child Welfare (MoHCW) declared that Zimbabwe would begin implementing Option B+ in October of 2013. This impact evaluation utilizes serial population-based, community-level surveys to comprehensively assess the prevention of mother-to-child HIV transmission strategy (PMTCT) 'Option B+' among mother-infant pairs in Zimbabwe. The investigators will assess the population-level impact of Option B+ in Zimbabwe using serial community-based cross-sectional serosurveys with data from three time points: 2012 (pre-Option A standard of care), 2014 (post-Option A / pre-Option B+), and 2017 (post Option B+ implementation) in order to monitor population-level trends in MTCT and HIV-free infant survival.

The investigators will compare outcomes among infants from 2017 to outcomes among mother-infant pairs who participated in similar surveys conducted in 2012 and 2014. These community-level data, along with in-depth facility survey data, will also allow the investigators to examine impact heterogeneity by the extent of integration of PMTCT and ART services at the facility. Together with effectiveness data from the serosurveys, facility-level resource utilization and cost data will allow assessment of Option B+ cost-effectiveness. In addition, this study will also include a population-based, community-level survey conducted in 2017 to assess retention of mothers in ART services after weaning (19-36 months postpartum). These data will allow the investigators to assess HIV-infected mothers' retention in care at the time of the survey, when most mothers will have stopped breastfeeding

ELIGIBILITY:
Inclusion Criteria Mothers-Infant pairs:

* Mother or caregiver is 16 years of age or older
* Delivered or provides care for an infant (alive or deceased) who is or who would have been 9-18 months of age at the time of the survey
* Able and willing to provide written informed consent

Exclusion Criteria Mothers-Infant pairs:

* Mother or caregiver is younger than 16 years of age
* Infant (alive or deceased) is not/would not have been 9-18 months of age at the time of the survey

Inclusion Criteria Mothers/Caregivers:

* At least 16 years of age or older
* Delivered an infant (alive or deceased) who is or who would have been 19-36 months of age at the time of the survey
* Able and willing to provide written informed consent

Exclusion Criteria Mothers/Caregivers:

* Mother or caregiver is younger than 16 years of age
* Infant (alive or deceased) is not/would not have been 19-36 months of age at the time of the survey

Inclusion Criteria Healthcare Staff:

* At least 18 years of age or older
* Currently providing PMTCT services at one of the 157 selected facilities
* Able and willing to provide written informed consent

Exclusion Criteria Healthcare Staff:

* Health care staff is younger than 18 years of age
* Health care staff is not currently providing PMTCT services at one of the 157 selected facilities

Inclusion Criteria Providers:

* At least 18 years of age or older
* Currently providing ANC or ART care directly to clients at one of the 20 purposefully selected facilities
* Splitting time as a provider between one or more of the following HIV services: HIV testing and counseling (HTC), prevention of mother-to-child transmission (PMTCT), and male circumcision (MC)
* Able and willing to provide written informed consent

Exclusion Criteria Providers:

* Provider is younger than 18 years of age
* Currently not providing ART care directly to clients at one of the 20 purposefully selected facilities
* Does not split time as a provider between one or more of the following HIV services: HIV testing and counseling (HTC), prevention of mother-to-child HIV transmission (PMTCT), and male circumcision (MC)

Inclusion Criteria Patients:

* At least 18 years of age or older
* Received HIV testing and counseling (HTC), prevention of mother-to-child HIV transmission (PMTCT), or male circumcision (MC) services at one of the 20 purposefully selected facilities on the day of the interview
* Able and willing to provide verbal consent

Exclusion Criteria Patients:

* Patient is younger than 18 years of age
* Did not receive HIV testing and counseling (HTC), prevention of mother-to-child HIV transmission (PMTCT), or male circumcision (MC) services at one of the 20 purposefully selected facilities on day of interview

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All study participants will be enrolled from 157 health facilities and health facility catchment areas in Harare, Mashonaland West, Mashonaland Central, Manicaland, and Matabeleland South provinces in Zimbabwe. In Zimbabwe, the catchment area of a health facility has a radius of approximately 10 km (allowing for variation due to geography).
  Healthcare staff, providers, and patients will be sampled from health facilities, while mother-infant pairs and mothers/caregivers will be sampled from health facility catchment areas.
Sampling Method: Probability Sample
Enrollment: 30642 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Vertical transmission of HIV infection | 9-18 months after birth
  Proportion of infants born to HIV-infected mothers who were HIV-infected
HIV-free survival among infants exposed to HIV | 9-18 months after birth
  Proportion of infants born to HIV-infected mothers who were alive and HIV-uninfected

SECONDARY OUTCOMES:
Retention of mothers in antiretroviral therapy services (ART) services after weaning | 19-36 months postpartum
  The proportion of HIV-infected mothers who were initiated on ART and who continued ART after weaning
Time between weaning and discontinuation of antiretroviral therapy services (ART) among mothers who did not continue ART after weaning | 19-36 months postpartum
  Average time between delivery and discontinuation of ART among those mothers who did not continue ART
Heterogeneity of the impact of Option B+ on HIV-free survival among infants 9-18 months of age by the extent of integration of PMTCT and anti-retroviral therapy (ART) services at health facilities | Baseline
  HIV-free survival in health facility catchment areas stratified by the extent of integration of PMTCT and ART services at the health facility
Heterogeneity of the impact of Option B+ on mother-to-child transmission of HIV (MTCT) among infants 9-18 months of age by the extent of integration of PMTCT and anti-retroviral therapy (ART) services at health facilities | Baseline
  MTCT in health facility catchment areas stratified by the extent of integration of PMTCT and ART services at the health facility
Cost-effectiveness of Option B+ compared to the standard of care before Option A | Baseline
  Facility costing data and HIV-free survival and MTCT in health facility catchment areas in 2012 compared to 2017
Cost-effectiveness of Option B+ compared to Option A | Baseline
  Facility costing data and HIV-free survival and MTCT in health facility catchment areas in 2012 compared to 2014
Variability in health facility accesibility | Baseline
  Accessibility of health facilities assessed using exit interviews with patients receiving care at health facilities
Variability in health facility quality of available services | Baseline
  Quality of available services at health facilities assessed using exit interviews with patients receiving care at health facilities, and clinical vignettes and time and motion studies with healthcare providers at health facilities
Variability in health facility appropriateness of available services | Baseline
  Appropriateness of available HIV testing and counseling (HTC), prevention of mother-to-child transmission of HIV (PMTCT) and male circumcision (MC) services assessed using clinical vignettes with healthcare providers at health facilities

CONTACTS AND LOCATIONS:
Overall Officials: Frances Cowan, MSc, MD, Principal Investigator — Liverpool School of Tropical Medicine, The Centre for Sexual Health and HIV/AIDS Research Zimbabwe; Nancy Padian, MPH, Ph.D, Principal Investigator — University of California, Berkeley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koyuncu A, Dufour MK, McCoy SI, Bautista-Arredondo S, Buzdugan R, Watadzaushe C, Dirawo J, Mushavi A, Mahomva A, Cowan F, Padian N. Protocol for the evaluation of the population-level impact of Zimbabwe's prevention of mother-to-child HIV transmission program option B+: a community based serial cross-sectional study. BMC Pregnancy Childbirth. 2019 Jan 8;19(1):15. doi: 10.1186/s12884-018-2146-x. PMID 30621615